CLINICAL TRIAL: NCT02968953
Title: Treatment With UX007 (Triheptanoin) for a Single Patient (ERS) With Glucose Transporter 1 (GLUT1) Deficiency Syndrome
Brief Title: Treatment With UX007 for a Single Patient With GLUT1 Deficiency Syndrome
Status: No longer available | Type: Expanded Access
Sponsor: Jerry Vockley, MD, PhD (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor-Investigator, Jerry Vockley, MD, PhD, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: PRO16060524
Record Dates: First submitted 2016-11-16; First posted 2016-11-21 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Glucose Transporter 1 Deficiency Syndrome
MeSH Terms: interventions — triheptanoin

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Triheptanoin — A single patient with Glucose Transporter 1 (GLUT1) Deficiency Syndrome will receive tripheptanoin (UX007).
  Other Names: UX007

SUMMARY:
This treatment plan is intended for the use of UX007 (triheptanoin) in the treatment of a single patient with Glucose Transporter 1 (GLUT1) Deficiency Syndrome.

DETAILED DESCRIPTION:
This treatment plan is intended for the use of UX007 (triheptanoin) in the treatment of a single patient with Glucose Transporter 1 (GLUT1) Deficiency Syndrome. Patient has already tried the other acceptable treatments for GLUT1 with either side effects that caused treatment to be discontinued (Ketogenic Diet) or a current treatment that is not showing any efficacy and is difficult to sustain for a long duration given this patient's age (modified Atkins diet). Due to the patient's ongoing neuroregression and lack of other viable treatments, the use of UX007 (triheptanoin) is warranted. There is no comparable or satisfactory alternative therapy to treat this patient's severely debilitating condition and the potential benefits to the patient justify the potential risks of the treatment. The potential risks from UX007 (triheptanoin) are not unreasonable given the context of this patient's condition.

ELIGIBILITY:
Inclusion Criteria:

* This treatment plan is intended for the use of UX007 (triheptanoin) in the treatment of a single patient with Glucose Transporter 1 (GLUT1) Deficiency Syndrome.

Exclusion Criteria:

* Not applicable as study only includes one patient.

Min Age: 3 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Vockley, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Pascual JM, Liu P, Mao D, Kelly DI, Hernandez A, Sheng M, Good LB, Ma Q, Marin-Valencia I, Zhang X, Park JY, Hynan LS, Stavinoha P, Roe CR, Lu H. Triheptanoin for glucose transporter type I deficiency (G1D): modulation of human ictogenesis, cerebral metabolic rate, and cognitive indices by a food supplement. JAMA Neurol. 2014 Oct;71(10):1255-65. doi: 10.1001/jamaneurol.2014.1584. PMID 25110966
- [Background] Blumenschine M, Montes J, Rao AK, Engelstad K, De Vivo DC. Analysis of Gait Disturbance in Glut 1 Deficiency Syndrome. J Child Neurol. 2016 Nov;31(13):1483-1488. doi: 10.1177/0883073816661662. Epub 2016 Aug 10. PMID 27511993
- [Background] Mochel F, Hainque E, Gras D, Adanyeguh IM, Caillet S, Heron B, Roubertie A, Kaphan E, Valabregue R, Rinaldi D, Vuillaumier S, Schiffmann R, Ottolenghi C, Hogrel JY, Servais L, Roze E. Triheptanoin dramatically reduces paroxysmal motor disorder in patients with GLUT1 deficiency. J Neurol Neurosurg Psychiatry. 2016 May;87(5):550-3. doi: 10.1136/jnnp-2015-311475. Epub 2015 Nov 3. PMID 26536893